CLINICAL TRIAL: NCT06399744
Title: Role of Sclerotherapy in Treatment of Non-neoplastic Ovarian Cyst
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Asmaa Ahmed Syed Ahmed, Resident Doctor, Al-Azhar University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sclerotherapy
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2022-10

CONDITIONS: Benign Ovarian Cyst
Keywords: sclerotherapy; cyst aspiration; non-neoplastic ovarian cysts
MeSH Terms: interventions — Sclerotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trans-abdominal group (Other)
  Interventions: Procedure: sclerotherapy
- trans-vaginal group (Other)
  Interventions: Procedure: sclerotherapy

INTERVENTIONS:
Procedure: sclerotherapy — injection of sclerosing agent (tetracycline or polidocanol) into ovarian cyst after aspiration of its contents

SUMMARY:
The aim of this study was to evaluate the role of sclerotherapy (injection of tetracycline or injection of Polidocanol - 95% hydroxypolyethoxydodecane and 5% ethanol -) in treatment of non-neoplastic ovarian cysts by, percutaneous trans-abdominal approach or trans-vaginal approach.

DETAILED DESCRIPTION:
Ovarian cysts are fluid-filled sacs that form in or on an ovary. Such cysts are relatively common. Most are non-cancerous (benign) and disappear on their own. Ovarian cancer is more likely to occur in women over 50.

Most of the patients with ovarian cyst are symptomless and resolves spontaneously. If untreated, complications such as rupture, torsion, malignant transformation may occur.

Cyst rupture can lead to peritoneal signs, abdominal distension and bleeding, irregularity of the menstrual cycle and abnormal vaginal bleeding, dull bilateral pelvic pain may result from the lutein cysts.

Until recent times, surgery in the form of laparotomy or laparoscopy has been the first choice. However, ultrasonography guided aspiration of the cysts as an alternative treatment is the fast catching up and may even be procedure of choice in the management of ovarian cysts in a selected group of women as it has low recurrence rate, low risk, less cost and in most cases no hospital stay.

There are various types of ovarian cysts, such as functional cysts, follicular cysts, corpus luteum cysts, hemorrhagic cysts, theca-lutein cysts, peritoneal inclusion cysts or pseudo-cysts, polycystic ovaries and endometriomas.

Functional cysts do not regress when treated with combined oral contraceptives that they do with expectant management.

Ovarian cysts are common, affecting 20% of women at some point in their lives . Unlike unilocular cysts including septations, solid irregular wall, or internal plaques, the simple ovarian cyst is defined as an anechoic round or oval lesion. The maximum diameter of simple ovarian cysts in premenopausal women is less than 5 cm, they often disappear during the menstrual cycle and do not require further intervention. Larger cysts (5-7 cm) should be followed using ultrasonography. Cysts larger than 7 cm may require advanced imaging or surgery.

Differential diagnosis in the management of an adnexal mass is complex because of the scope of the disorders that may have caused it and the numerous therapies that may be appropriate. It is the risk of malignancy that propels protocols and procedures, as well as the fundamental concept that early diagnosis and treatment in cancer are related to lesser mortality and morbidity. Non neoplastic ovarian cysts in women with menstrual cycles are the most frequently detected masses involving the adnexa. Many of these cysts are functional and resolve spontaneously within a few days to 2 weeks, but they can persist longer.

The management of women with benign ovarian cysts remains controversial. Various treatment protocols use medical treatment (mainly oral contraceptives), ultrasound-guided aspiration, laparoscopy (cystectomy or drainage and ablation of the cystic wall) and laparotomy (cystectomy) Sclerotherapy of ovarian cysts has been attempted to decrease the probability of recurrence. Although ultrasound-guided aspiration is simple and safe, the recurrence rate is high, ranging from 28.5% to 100%. In order to reduce this rate, ultrasound-guided ethanol sclerotherapy for ovarian cysts was first introduced in 1988, and it has been reported by several authors to be simple and safe.

Tetracycline, methotrexate, and ethanol are the most common agents used for sclerotherapy. When compared to women without cysts, sclerotherapy applied to infertile women with ovarian cysts has been shown to reduce pelvic pain without affecting the number of follicles, term pregnancy and abortion rates, the number of obtained oocytes, embryo quality, or hormonal levels.

We chose either tetracycline or Polidocanol as sclerosing agents. Tetracycline because of its antibacterial effect, which may help to control infections. Tetracyclines (tetracycline, doxycycline, minocycline) have been used as sclerosing agent in various clinical settings such as pleural effusions, pneumothoraxes, hydroceles, benign lymphoepithelial cysts of the parotid gland and lymphoceles after renal transplantation.

Polidocanol is a nonionic surfactant sclerosing agent, which consists of 95% hydroxypolyethoxydodecane and 5% ethanol. Polidocanol was invented as an anesthetic agent. Polidocanol is a liquid surfactant having endothelial cell lytic properties.

The mechanism underlying the sclerosing effect was generally attributed to the results of local chemical irritation or inflammatory response. Ethanol induces a combination of cytotoxic damage, dehydration of cells, and production of mediators for inflammation and fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients were diagnosed with non-neoplastic ovarian cysts (i.e., simple, hemorrhagic, complicated, endometriotic cysts).
* All Patients from 15 to 48 years old.
* Size from (5 to 10 cm).
* Cyst wall thickness < 5 mm.
* Negative tumor markers (Cancr Antigen125, Cancer Embryonic Antigen, Cancer Antigen19.9 & alpha fetoprotein).
* Persisted for more than 3 months.
* Normal color Doppler blood flow analysis.
* Resistant to hormonal treatment COCs.
* Patients accepted to be enrolled in the study.

Exclusion Criteria:

* Family history of ovarian cancer.
* USG features suggesting malignancy like: multilocular, papillary projections or mural nodule, cyst wall thickness >5mm, low Doppler indices (PI≤1 and or RI≤0.40, centrally located vessels, randomly dispersed vessels).
* Known allergy to sclerosing agent (tetracycline or Polidocanol).
* Bleeding tendency as (patients with platelet count <50,000, patients with Uncorrected Coagulopathy with International Normalized Ratio >1.5, or patients on antithrombotic therapy without stoppage of doses till 5 days before the procedure.

Ages: 15 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
role of sclerotherapy in treatment of non-neoplastic ovarian cysts | followed up from 1 month to 6 months
  The main outcome measure was the disappearance of the cyst and the avoidance of surgery. The cyst was considered resolved if follow-up revealed either no cystic lesion or only a follicle-like cyst no more than 30 mm in diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Abdallah, Study Director — Al-Azhar University
Locations (1):
- Al-Azhar University, Asyut, Egypt